CLINICAL TRIAL: NCT04721002
Title: MEDICI - t(11;14) and BCL2 Expression in Patients With Multiple Myeloma: Prevalence, Stability Across Lines of Therapy and Concordance Across Sample Types
Brief Title: Study to Evaluate t(11;14) Status and BCL2 Expression in Adult Participants With Multiple Myeloma (MM)
Acronym: MEDICI
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: H20-126
Record Dates: First submitted 2021-01-21; First posted 2021-01-22 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Multiple Myeloma (MM)
Keywords: Multiple myeloma (MM); Relapsed/Refractory (R/R) Multiple myeloma (MM); t(11; 14); BCL2
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone marrow aspirate and peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants With Multiple Myeloma: Participants with newly diagnosed and relapsed/refractory multiple myeloma will receive standard of care. Bone marrow and blood samples will be collected.

SUMMARY:
Multiple myeloma (MM) is a rare cancer caused by abnormal survival of plasma cells (blood cells). Most trial participants with MM relapse (cancer has come back) or become non- responsive to treatment and remission gets shorter after each line of treatment. This is a study to assess t(11;14) and BCL2 expression in adult participants with newly diagnosed and relapsed/refractory (R/R) MM.

Approximately 500 adult participants with newly confirmed or relapsed/refractory (R/R) multiple myeloma (MM) will be enrolled in around 15-20 countries.

Participants will receive standard of care while participating in this study. No drug will be administered as a part of this study.

Participants will attend regular visits during the course of the study at a hospital or clinic and will be asked to provide bone marrow and blood samples.

ELIGIBILITY:
Inclusion Criteria:

- Confirmed newly diagnosed or relapsed/refractory (R/R) Multiple myeloma (MM) who have signed informed consent for the use of their biological material for research purposes.

Exclusion Criteria:

- Participants who do not have Bone Marrow (BM) and blood sample at time of diagnosis or at confirmation of relapse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with confirmed newly diagnosed or relapsed/refractory multiple myeloma
Sampling Method: Non-Probability Sample
Enrollment: 514 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With t(11;14) Status by Fluorescence In Situ Hybridization (FISH) Analysis of Bone Marrow Plasma Cells | Up to approximately 2.5 months following last subject last visit
  t(11;14) status (positive or negative) of the earliest multiple myeloma (MM) sample collected at initial diagnosis or across lines of therapies, by FISH analysis of bone marrow plasma cells is evaluated.
Percentage of Participants With BCL2 Status by Quantitative Polymerase Chain Reaction (qPCR) Analysis of Bone Marrow Plasma Cells | Up to approximately 2.5 months following last subject last visit
  BCL2 status (BCL2 high or not) of the earliest MM sample collected, either at initial diagnosis or across lines of therapies, by qPCR analysis of bone marrow plasma cells is evaluated.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Stability of t(11;14) Status | Up to approximately 2.5 months following last subject last visit
  Stability of t(11;14) status across intra-patient longitudinal bone marrow (BM) samples (changed vs not changed) collected at initial diagnosis and across lines of therapies.
Percentage of Participants Achieving Stability of BCL2 Status | Up to approximately 2.5 months following last subject last visit
  Stability of BCL2 status across intra-patient longitudinal BM samples (changed vs not changed) collected at initial diagnosis and across lines of therapies.
Percentage of Participants With t(11;14) Status Determined by Bone Marrow (BM) Biopsy | Up to approximately 2.5 months following last subject last visit
  t(11;14) status (positive or negative) at initial diagnosis and across lines of therapy as determined by BM biopsy.
Percentage of Participants With BCL2 Status Determined by Bone Marrow Biopsy | Up to approximately 2.5 months following last subject last visit
  BCL2 status (BCL2high or BCL2low) at initial diagnosis and across lines of therapy as determined by BM biopsy.
Percentage of Participants With t(11;14) Status of MM Samples | Up to approximately 2.5 months following last subject last visit
  t(11;14) status (positive or negative) of MM samples at different disease stages as determined by BM biopsy.
Percentage of Participants With BCL2 Status of MM Samples | Up to approximately 2.5 months following last subject last visit
  BCL2 status (BCL2high or BCL2low) of MM samples at different disease stages as determined by BM biopsy.
Percentage of Participants With t(11;14) Status of MM Samples at Different Treatment Lines Stages | Up to approximately 2.5 months following last subject last visit
  t(11;14) status (positive or negative) of MM samples at different treatment lines stages as determined by BM biopsy.
Percentage of Participants With BCL2 Status of MM Samples at Different Treatment Lines Stages | Up to approximately 2.5 months following last subject last visit
  BCL2 status (BCL2high or BCL2low) status of MM samples at different treatment lines stages as determined by BM biopsy.
Percentage of Participants With t(1;14) Status and BCL2 Status | Up to approximately 2.5 months following last subject last visit
  t(11;14) and BCL2 status (Positive and BCL2high, Negative and BCL2high, Positive and BCL2low, Negative and BCL2low) of the earliest MM samples collected, at initial diagnosis or across lines of therapies, by FISH and qPCR analyses of bone marrow plasma cells, respectively.
Percentage of Participants With FISH Fusion (F) Categories as Determined by BM Biopsy | Up to approximately 2.5 months following last subject last visit
  FISH fusion (F) categories (1F, 2F, >=3F) among t(11;14) positive samples as determined by BM biopsy.
Percentage of Participants With FISH Fusion (F) Categories Across Lines of Therapies as Determined by BM Biopsy | Up to approximately 2.5 months following last subject last visit
  FISH fusion (F) categories (1F, 2F, >=3F) among t(11;14) positive samples across lines of therapies as determined by BM biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (40):
- United States (2):
  - Tulane School of Medicine /ID# 223864, New Orleans, Louisiana
  - University of Texas Southwestern Medical Center /ID# 223865, Dallas, Texas
- Hospital Italiano de Buenos Aires /ID# 224153, Ciudad Autonoma Buenos Aires, Buenos Aires F.D., Argentina
- Alfred Health /ID# 224386, Melbourne, Victoria, Australia
- Brazil (7):
  - Hospital São Rafael /ID# 224307, Salvador, Estado de Bahia
  - Hospital de Clinicas de Porto Alegre /ID# 224274, Porto Alegre, Rio Grande do Sul
  - Clinica Sao Germano /ID# 224239, São Paulo, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein /ID# 224303, São Paulo, São Paulo
  - Instituto COI de Educacao e Pesquisa /ID# 224245, Rio de Janeiro
  - Real e Benemérita Associação Portuguesa de Beneficência /ID# 224305, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo /ID# 225749, São Paulo
- Cross Cancer Institute /ID# 224172, Edmonton, Alberta, Canada
- Klinicki bolnicki centar Zagreb /ID# 226969, Zagreb, City of Zagreb, Croatia
- Czechia (2):
  - Fakultni nemocnice Hradec Kralove /ID# 224089, Hradec Králové
  - Fakultni nemocnice Ostrava /ID# 224090, Ostrava
- France (3):
  - CHRU Lille - Hopital Claude Huriez /ID# 228919, Lille, Hauts-de-France
  - CHU de Nantes, Hotel Dieu -HME /ID# 223702, Nantes, Pays de la Loire Region
  - AP-HP - Hopital Necker /ID# 228062, Paris
- Germany (2):
  - Praxis am Volkspark /ID# 224763, Berlin
  - Asklepios Klinik Altona /ID# 224761, Hamburg
- Alexandra General Hospital /ID# 224828, Athens, Attica, Greece
- Beaumont Hospital /ID# 225514, Beaumont, Dublin, Ireland
- Hadassah Medical Center-Hebrew University /ID# 224884, Jerusalem, Jerusalem, Israel
- Italy (2):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona /ID# 224690, Ancona
  - ASST Grande Ospedale Metropolitano Niguarda /ID# 224608, Milan
- Maastricht Universitair Medisch Centrum /ID# 224694, Maastricht, Netherlands
- Rikshospitalet OUS HF /ID# 227288, Oslo, Norway
- Poland (2):
  - Szpital Kliniczny im. Heliodora Swiecickiego Uniwersytetu Medycznego im. Karola /ID# 227038, Poznan, Greater Poland Voivodeship
  - Instytut Hematologii i Transfuzjologii /ID# 227039, Warsaw, Masovian Voivodeship
- Institutul Clinic Fundeni /ID# 224574, Bucharest, București, Romania
- Princess Noorah Oncology Center /ID# 224968, Jeddah, Saudi Arabia
- Univ Medical Ctr Ljubljana /ID# 225408, Ljubljana, Slovenia
- Spain (6):
  - Hospital Universitario Germans Trias i Pujol /ID# 229281, Badalona, Barcelona
  - Hospital Clinic de Barcelona /ID# 224804, Barcelona
  - Hospital de Leon /ID# 229191, León
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 229524, Madrid
  - Hospital Universitario 12 de Octubre /ID# 225617, Madrid
  - Hospital Universitario de Salamanca /ID# 224803, Salamanca
- Taichung Veterans General Hospital /ID# 227084, Taichung, Taiwan
- Bagcilar Medipol Mega Universite Hastanesi /ID# 225515, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Spencer A, Gavriatopoulou M, Coriu D, Lysen A, Gutierrez NC, Escalante F, Eugenia Fantl DB, Hajek R, Seguro F, Kaur G, Bittencourt R, Kinda SB, Chu MP, Safah H, Martinez-Lopez J, de Queiroz Crusoe E, Cordeiro de Farias DL, Offidani M, Askari E, Sevindik OG, Maisnar V, Teng CL, Hughes O, Taylor R, Lehn K, Feng D, Thiebaut-Millot R, Li X, Murray L, Jung P, Rossi EL, Kongpachith S, Nichol A, Ross JA, Hader C. Prospective real-world evaluation of t(11;14) prevalence and disease biology in multiple myeloma: MEDICI study analysis. Blood Adv. 2025 Nov 25;9(22):5814-5827. doi: 10.1182/bloodadvances.2025017214. PMID 40829119